CLINICAL TRIAL: NCT02582983
Title: An Open-Label Safety Trial of Enfuvirtide (T-20/RO 29-9800, HIV-1 Fusion Inhibitor) in Combination With Free Choice Antiviral Regimen in Thai Patients With Advanced HIV Infection
Brief Title: A Study of Enfuvirtide (Fuzeon) in Participants With Advanced Human Immunodeficiency Virus (HIV) Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML17819
Record Dates: First submitted 2015-10-08; First posted 2015-10-21 (Estimated); Results first posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

ARMS (1):
- Enfuvirtide (Experimental): Participants received Enfuvirtide 90 mg subcutaneously (SC) twice daily (BID).
  Interventions: Drug: Enfuvirtide

INTERVENTIONS:
Drug: Enfuvirtide — All participants received enfuvirtide 90 mg SC BID until 4 weeks after commercial availability was established in Thailand.
  Other Names: Fuzeon

SUMMARY:
This study assessed the safety and tolerability of enfuvirtide in participants with advanced HIV genotype 1 (HIV-1) disease. Eligible participants who failed treatment with regimens containing at least one product from each anti-retroviral class, or had experienced intolerance to previous anti-retroviral regimens received enfuvirtide, 90 milligrams (mg) subcutaneously (SC) twice daily (BID) as long as there were no enfuvirtide related treatment limiting toxicities and participants benefited from study treatment as per investigator's discretion. The anticipated time on study treatment was based on the commercial availability of enfuvirtide in Thailand, and the target sample size was 30 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals at least 16 years of age infected with HIV-1
* CD4 lymphocyte count less than equal to (<=) 100 cells per cubic millimeter (cells/mm^3) and HIV-1 ribonucleic acid (RNA) viral load greater than equal to (>=) 10,000 copies/mL while on highly active antiretroviral therapy (HAART)
* Genotypic or phenotypic resistance and/or treatment-limiting toxicity on previous antiretroviral regimens

Exclusion Criteria:

* Evidence of ongoing alcohol and/or drug or substance abuse
* Prior non-adherence to antiretroviral treatment regimens
* Evidence of active, untreated opportunistic infection, intercurrent illness, drug toxicity or any other condition.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (3):
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Nonthaburi

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enfuvirtide
Started | 23
Completed | 17
Not Completed | 6
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Enfuvirtide
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.17 (8.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A serious adverse event is any untoward medical occurrence that at any dose: results in death, or is life-threatening, or requires inpatient hospitalization or prolongation of existing hospitalization, or results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect. The term "life-threatening" in the definition of "serious" refers to an event in which the patient was at risk of death at the time of the event, not an event which hypothetically might have caused death if it were more severe.
Time Frame: Up to 28 days after permanent discontinuation of study treatment (approximately 100 weeks)
Population: The analysis population was defined as the number of participants who enrolled in the study and received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Enfuvirtide
Number analyzed (Participants) | 23
participants | 6

2. Primary Outcome: Number of Participants With Premature Withdrawal Due to Adverse Events
Time Frame: Up to 96 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Enfuvirtide
Number analyzed (Participants) | 23
participants | 1

ADVERSE EVENTS:
Time Frame: Up to 28 days after permanent discontinuation of study treatment (approximately 100 weeks)
Arm/Group | Enfuvirtide
Serious Adverse Events (participants affected / at risk) | 6/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enfuvirtide (N=23)
Anaemia (Blood and lymphatic system disorders) | 1
Cellulitis (Infections and infestations) | 2
Pancreatitis acute (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Immune reconstitution inflammatory syndrome (Immune system disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Headache (Nervous system disorders) | 1
Brain stem stroke (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enfuvirtide (N=23)
Injection site pain (General disorders) | 14
Injection site induration (General disorders) | 13
Injection site reaction (General disorders) | 5
Injection site haemorrhage (General disorders) | 6
Injection site rash (General disorders) | 5
Injection site oedema (General disorders) | 4
Injection site erythema (General disorders) | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 8
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 6
Cytomegalovirus infection (Infections and infestations) | 3
Anorexia nervosa (Psychiatric disorders) | 2
Pyrexia (General disorders) | 2
Congenital herpes simplex infection (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 2
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Cold (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.